CLINICAL TRIAL: NCT06750822
Title: Accuracy of Automatic Contusion Volume Scanning for Predicting the Incidence of Pneumonia in Patients With Thoracic Trauma
Acronym: RESOLUTION
Status: Completed | Type: Observational
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Other Study IDs: 24057-667-2024-OSS-RESOLUTION
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pneumonia; Thoracic Trauma
Keywords: AAST; AISThorax; Pneumonia; trauma
MeSH Terms: conditions — Pneumonia; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma patients: Any patient admitted for trauma in the Emergency Department receiving a whole-body contrast CT scan.

SUMMARY:
The goal of this retrospective observational study is to evaluate the diagnostic accuracy of pulmonary contusion volume in predicting early pneumonia in patients with thoracic trauma.

The primary question we aim to answer is: What is the diagnostic accuracy of pulmonary contusion volume in predicting pneumonia within 7 days post-trauma?

Moreover, we aim to explore which is the overlap between the contused segments and those developing pneumonia.

Finally, we aim to explore relevant differences in radiomic features between contused segments that developed pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the ED for trauma as primary diagnosis
* Whole-body contrast CT scan performed within 6 hours from admission

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes all the consecutive patients admitted to the ED of the institution for trauma and having a contrast whole-body CT scan performed within 6 hours from admission
Sampling Method: Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
7d-pneumonia | 7 days
  Pneumonia appearing within 7 days from trauma, defined as:
  • New or worsening pulmonary infiltrates plus ≥ 2 of the following:
  * Body temperature ≥ 38°C or ≤ 35°C
  * White Blood Cell (WBC) count > 12,000 or < 4,000 cells/mL or presence of immature granulocytes in the blood sample
  * Purulent sputum
  * Worsening pulmonary oxygenation, defined as a decline in the PaO2/FiO2 ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Maggiore Hospital Carlo Alberto Pizzardi, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared upon reasonable request

REFERENCES:
- [Derived] Gamberini L, Astuti GM, Biavati B, Boarato D, Tontodonati M, Palmitessa I, Laruccia M, Coniglio C, Bertini A, Orlandi PE, Tartaglione M, Allegri D, Bruno A. Pulmonary contusion volume and radiomics as predictors of early-onset pneumonia in trauma patients, a retrospective single-centre study. Eur J Trauma Emerg Surg. 2025 Aug 22;51(1):275. doi: 10.1007/s00068-025-02952-1. PMID 40844714